CLINICAL TRIAL: NCT02883491
Title: Pulmonary Embolism Short-term Clinical Outcomes Registry (PE-SCOR)
Brief Title: Pulmonary Embolism Short-term Clinical Outcomes Registry
Acronym: PE-SCOR
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00082655; 07-16-06E (Other: Atrium)
Record Dates: First submitted 2016-08-19; First posted 2016-08-30 (Estimated); Last update posted 2022-04-26 (Actual); Status verified 2020-01

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overall goal of this clinical research study is to prospectively assess primary outcomes related to pulmonary embolism (PE) that occur immediately (within 5 days) and within 30 days. The secondary goal is to compare validated prediction models and a modified European Society of Cardiology (ESC) approach that is primarily right ventricle dysfunction (RVD) driven with clinical risk assessment being secondary, and with primary outcomes of clinical deterioration within 5 days.

DETAILED DESCRIPTION:
The investigators wish to develop the Pulmonary Embolism Short-term Clinical Outcomes Registry (PE-SCOR). The investigators also wish to determine the incidence of death and circulatory and respiratory deterioration, and administration of reperfusion therapy within 5 days in PE patients. The study will also evaluate the sensitivity, specificity and positive and negative predictive values of each RVD assessment option. The investigators will also derive a prediction model for PE patients for the primary outcome within five days. Finally, investigators will determine the functional outcomes of PE patients 30 days after PE.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older with image confirmed acute pulmonary embolism diagnosed within 12 hours of ED presentation will be eligible for enrollment.

Exclusion Criteria:

* Patients who refuse consent for 30-day clinical contact and follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who present to the Emergency Department (ED) with image confirmed acute pulmonary embolism diagnosed within 12 hours of presentation.
Sampling Method: Probability Sample
Enrollment: 815 (Actual)
Dates: Start 2016-08; Primary Completion 2019-02-20 (Actual); Study Completion 2019-02-20 (Actual)

PRIMARY OUTCOMES:
Clinical Deterioration | 5 days
  Presence of any one clinical deterioration variable: death, circulatory or respiratory dysfunction, reperfusion interventions.
Right ventricular dysfunction (RVD) | Index visit
  Presence of any one indicator of RVD: any one goal directed echocardiography finding of RVD (right ventricle (RV) enlargement or, leftward deviation of the interventricular septum, or RV systolic dysfunction by longitudinal movement of the tricuspid annulus of the RV free wall), CT right ventricle : left ventricle ratio greater or equal to 1, positive troponin or B-type Natriuretic Peptide, EKG injury and ischemia patterns of RVD

SECONDARY OUTCOMES:
Functional Outcome | 30 days
  Pulmonary Embolism Quality of Life (PEmb-QoL) questionnaire
Pulmonary Embolism Complications | 30 days
  Presence of any one variable: recurrence of pulmonary embolism, subsequent hospitalizations, major and minor bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Weekes, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (6):
- United States (6):
  - San Diego Medical Center, San Diego, California
  - Christiana Care Health System, Newark, Delaware
  - Orlando Regional Medical Center, Orlando, Florida
  - Carolinas Healthcare System, Charlotte, North Carolina
  - Vanderbilt Medical Center, Nashville, Tennessee
  - University of Utah Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No